CLINICAL TRIAL: NCT06507189
Title: Multidimensional Predictive Modeling to Understand Mechanisms of Exercise Response Heterogeneity in Older Adults
Brief Title: Multidimensional Predictive Modeling to Understand Mechanisms of Exercise Response Heterogeneity in Older Adults (M3AX)
Acronym: M3AX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Collaborators: University of Florida (Other); Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-0083
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The overarching goal of this project is to determine factors contributing to response heterogeneity in outcomes key to healthy aging. The first phase of this two-phase trial will be focused on understanding the underlying biological mechanisms that explain/predict response heterogeneity and the second phase will test augmentation efforts to mitigate poor responsiveness while assessing whether the same or different mechanisms predict response when augmenting an individual's prescription in Phase II.
Who Masked: Investigator
Masking Description: Biospecimen investigators will be blinded from gender and age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrogation (Experimental): In Interrogation, all participants will exercise train using an exercise prescription that is in accordance with current public health recommendations19. At the end of Phase I participants will be classified into one of the four categories listed in Fig. A: (1) CRF-/fMQ-, 2) CRF-/fMQ+, 3) CRF+/fMQ- and 4) CRF+/fMQ+).
  Interventions: Other: Combined endurance and resistance training
- Mitigation (Experimental): Based on these categories of responsiveness, exercise training will be boosted in the three groups that are nonresponsive in one or both outcomes. CRF-/fMQ+ will receive boosted ET, CRF+/fMQ- will receive boosted RT, and CRF-/fMQ- will receive boosting in both. All three of these classifications will also receive education on wearable device data and other free-living recommendations four times during Mitigation
  Interventions: Other: Combined endurance and resistance training

INTERVENTIONS:
Other: Combined endurance and resistance training — ET will consist of 3x/wk training (MWF) with MF being steady state cycling, treadmill, or elliptical at 70-75% HRR for 30 min and the W session being a 20 min high intensity interval session on a cycle ergometer (1 min on/off; 10 cycles) targeting 85-90% HRR. The treadmill and elliptical on M or F will be provided for variety but the mainstay will be cycle ergometry. On MF participants will complete 3 sets x 8-12 repetitions for leg press, knee extension, hamstring curl, chest press, seated row, overhead press, lat pulldown, triceps push-down, and biceps curl in superset fashion [i.e., alternate between opposing muscle groups without rest (chest press followed by seated row)] with a 60 s rest between supersets. Sets will be performed with load progression to ensure volitional fatigue in the 8-12 rep range. Core exercises (trunk flexion and extension) will also be included using bodyweight only for 3 sets.

SUMMARY:
Aging-related functional declines are thought to be caused by hallmark biological processes that ultimately manifest in physical, mental, and metabolic impairments that compromise healthspan and quality of life. Exercise is a multipotent treatment with promise to mitigate most aging hallmarks, but there is substantial variability in exercisƒe responsiveness. Combining endurance and resistance training in alignment with public health guidelines will be used to better understand variable exercise responsiveness in older adults with the ultimate goal of improving each older adult's capacity to attain the many health benefits of exercise.

DETAILED DESCRIPTION:
Aging-related functional declines are thought to be caused by hallmark biological processes1 that ultimately manifest in physical, mental, and metabolic impairments - compromising healthspan and quality of life (QoL). Exercise is a multipotent treatment with promise to mitigate most aging hallmarks, but there is substantial variability in individual exercise responsiveness. This inter-individual response heterogeneity (IRH) was first identified and extensively interrogated by Bouchard and colleagues in the context of endurance training (ET). Subsequently, the investigators have demonstrated resistance training (RT) IRH and have studied potential IRH mechanisms. The investigators then led multiple trials in older adults examining dose titration, adjuvant nutrition or medication in attempts to lower poor response rates. Many knowledge gaps remain as summarized in the National Institutes of Aging (NIA) workshop on IRH seeding this Requests for Applications (RFA). The investigators have assembled an interdisciplinary team to address the RFA's central goal, "to better understand factors underlying response variability to exercise training in older adults." Although Health and Human Services (HHS) guidelines specify combined ET and RT to maximize health benefits in aging adults, large-scale exercise trials studying IRH (i.e., HERITAGE, MoTrPAC) have restricted participants to a single exercise mode. For this project, the investigators propose the innovative, but logical, strategy to use combined ET and RT. Low cardiorespiratory fitness (CRF, VO2max) and low functional muscle quality (fMQ; strength/muscle mass) are multi-system manifestations of the deterioration of the cellular hallmarks of aging. Importantly, both CRF and fMQ are modifiable with ET and RT. Thus, the investigators design premise is that combined ET+RT is an excellent strategy for elucidating factors underlying IRH, as it forges a path toward understanding and mitigating IRH in aging with direct translatability to best-evidence public health recommendations.

It is yet to be determined how the hallmarks of aging interact to influence exercise responsiveness. For example, muscle mitochondrial energetics and proteostasis are inextricably linked, and poor responder status may be caused by lack of energetic resources to maintain proteostasis throughout an exercise program. Similarly, aging disrupts circadian clocks, leading to inflammation and disrupted cell signaling, which may also contribute to IRH.

While sources of IRH are a constellation of modifiable and non-modifiable factors, the investigators will test the hypothesis that factors central to aging itself - aging hallmarks such as proteostasis, mitochondrial energetics, and inflammation, as well as systemic and muscle-specific circadian clock function and output - are chief contributors to the multidimensional circuitry that determines whether an individual achieves the minimum clinically important difference (MCID) in CRF and/or fMQ with exercise training. The investigators will also test the hypothesis that altered exercise dosing coupled with lifestyle recommendations will promote attainment of MCIDs among older adults who do not initially respond. With CRF and fMQ as primary clinical outcomes, the investigators will use a 2-phase Sequential Multiple Assignment Randomized Trial (SMART) of combined ET+RT with clinical phenotyping and blood/muscle molecular and cellular analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 60 or above
2. Free of chronic disease
3. No structured exercise program (2 or more bouts/wk) within previous 12 months
4. Cognitively capable of providing informed consent

Exclusion Criteria:

1. Neuromuscular or musculoskeletal disorder that would limit ability to perform the exercise and/or testing bouts
2. Cardiopulmonary disorders or reduced breathing capacity (FEV1 < 80% expected)
3. Metabolic diseases including markers of liver disease (ALT > 52 U/l) and type 2 diabetes (HbA1C ≥ 6.5, fasting blood glucose ≥ 126 mg/dl)
4. Any other disease or disorder that would influence exercise response (e.g., chronic kidney disease, dementia, current cancer diagnosis or within 2 yr remission, cerebrovascular disease)
5. Any current infectious disease
6. Life expectancy < 1 year
7. Insulin sensitizing/blood glucose lowering agents such as metformin
8. High dose lipophilic statin (≥40 mg/d)
9. Lidocaine allergy
10. Regular tobacco use and/or vaping
11. Excessive alcohol consumption (3 drinks/d or 7 drinks/wk for females; 4 drinks/d or 14 drinks/wk for males)
12. BMI ≥ 30.0 kg/m2
13. Unable to commit to ~6 months required to complete the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (CRF) | 23 weeks
  A primary outcome of this investigation is cardiorespiratory fitness (CRF). The CRF is the amount of oxygen (ml/kg) that is used during exercise and how efficient you are using that oxygen. The exercise used to measure oxygen uptake is a stationary bicycle with increasing intensity until you are able to maintain pace. Your expired air is collected with a mask or mouthpiece and analyzed with an oxygen and carbon dioxide sensor.
Functional muscle quality (fMQ) | 23 weeks
  A primary outcome of this investigation is functional muscle quality (fMQ). This is a ratio of knee extension strength to thigh leanness. Knee extension strength is the maximum amount of weight you can successfully lift one time. Thigh lean mass is measured with the dual energy x-ray absorptiometry (DEXA). This is a common tool used to measure bone density, but it is very efficient at determining fat and lean masses partitioned in the body.

SECONDARY OUTCOMES:
Balance | 23 weeks
  Balance will be assessed with tools such at the short physical performance battery (SPPB). The SPPB is a clinical test used to measure balance in three areas of balance: stand-in balance, gait speed and chair stand time. The overall higher score you have is an indicator of better balance.
Cognitive performance | 23 weeks
  An assessment such as the Trail Making Task (TMT)is used to measure reaction times at the beginning of and after the exercise intervention.
Body composition | 23 weeks
  Body composition will be measured four times pre and post to exercise intervention.
Metabolic health | 23 weeks
  A clinical assessment such as continuous glucose monitoring (CGM) will be use to measure metabolic health at the beginning, the middle, and end of intervention time points. CGM will monitored for seven days pre and post to the exercise intervention. This can be used to determine blood glucose response before and after exercise.
Metabolic health | 23 weeks
  The HOMA-IR will is test used to determine protein turn over or how efficient you are at processing proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Marcas Bamman, Principal Investigator — Florida Institute for Human and Machine Cognition
Locations (2):
- United States (2):
  - Florida Institute for Human and Machine Cognition, Pensacola, Florida
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
Data Entry and Management System. Regarding the data entry and management system (DEMS) used for data management, we will customize one of the DEMS platforms developed by the team at IHMC using Smartabase, which is a federally approved, secure cloud-based environment we are currently using in other federally funded observational studies and clinical trials. We have experienced Smartabase builders on the team led by Dr. McAdam who will create custom programs and forms for the study that facilitate data collection and entry while also having the infrastructure to provide access to real-time data summaries and comparisons across all performance sites. Importantly, we have established numerous streamlined approaches for direct electronic data transfer to Smartabase from testing instruments (e.g., DXA, metabolic carts, strength dynamometers, EMG systems) via APIs to eliminate manual data entry errors.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be transferred and monitored on the day of acquisition. Data will be identified with unique study identity.